CLINICAL TRIAL: NCT01225666
Title: A Phase II, Dose and Frequency Finding Study of MOD-4023 in Growth Hormone Deficient Adults (GHDA)
Brief Title: MOD-4023 (Long-Lasting Human Growth Hormone (hGH)) Study in Growth Hormone Deficient Adults (GHDA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-4-003; 2010-019374-32 (EudraCT Number)
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Adult Growth Hormone Deficiency
Keywords: MOD-4023; Growth Hormone Deficient Adults; Phase II
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — MOD-4023

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Weekly low dose (Experimental): MOD-4023
  Interventions: Drug: MOD-4023
- Weekly middle dose (Experimental): MOD-4023
  Interventions: Drug: MOD-4023
- Weekly high dose (Experimental): MOD-4023
  Interventions: Drug: MOD-4023
- Every-other week dose (Experimental): MOD-4023
  Interventions: Drug: MOD-4023

INTERVENTIONS:
Drug: MOD-4023 — liquid solution for subcutaneous injection - 30% of the cumulative weekly dose achieved with daily rhGH, Once weekly
  Arms: Weekly low dose
Drug: MOD-4023 — liquid solution for subcutaneous injection - 45% of the cumulative weekly dose achieved with daily rhGH, Once weekly
  Arms: Weekly middle dose
Drug: MOD-4023 — liquid solution for subcutaneous injection - 100% of the cumulative weekly dose achieved with daily rhGH, Once weekly
  Arms: Weekly high dose
Drug: MOD-4023 — liquid solution for subcutaneous injection - 100% of the cumulative weekly dose achieved with daily rhGH, every-other week (50% of the two-weekly cumulative dose)
  Arms: Every-other week dose

SUMMARY:
This study aims to assess the safety, tolerability and Pharmacokinetics/ Pharmacodynamics (PK/PD) profile of three doses of MOD-4023 on a weekly regime and one dose on an every-other-week regime administered for a period of 4 weeks in Growth Hormone Deficient Adult (GHDA) patients who previously were on a stable r-hGH treatment. An additional extension period of 16 weeks once-weekly administration of MOD-4023 aims to confirm the dose selection for future trials.

DETAILED DESCRIPTION:
The study is a phase II, randomized, open-label, parallel, 4 active treatment arms study to evaluate the safety, tolerability and PK/PD profile of MOD-4023 in pre-treated, normalized, GHD adults.

The study is conducted in 2 stages. Stage I is a 4-week treatment period with 4 different dose levels/dosing regimens.

Stage II is a 16-week treatment-extension period in which all the patients will start with the same dose (derived from stage I) and will be dose titrated to maintain IGF-1 levels within the normal range.

ELIGIBILITY:
Inclusion Criteria:

* Genders Eligible for Study: Both
* Ages Eligible for Study: Males - 23 to 60 years, Females - 23 to 50 years.
* GHDA subjects as defined in the Consensus guidelines for the diagnosis and treatment of adults with GH deficiency II (2007).
* Patients using hormonal replacement therapy(s) for deficiencies of other hypothalamo-pituitary axes must be on an optimized and stable treatment regimen (hormone levels within normal ranges on screening) for at least three months prior to screening:

  * Temporary adjustment of glucocorticoid replacement therapy, as appropriate, is acceptable.
  * Peripheral thyroid hormones (FT4, FT3) within the normal range.
* Fertile females must agree to use appropriate contraceptive methods
* Female patients must have a negative serum pregnancy test at inclusion.
* Growth Hormone (GH) replacement therapy for more than 6 months with registered GH product.
* The IGF-I level at screening within -1.5 to +1.5 SDS of the age and sex normal ranges according to the central laboratory measurements.
* Body Mass Index (BMI, kg/m2) of 22.0 to 35.0 kg/m2, both inclusive
* Confirmed to be negative for anti r-hGH antibodies at the time of screening.
* Willing and able to provide written informed consent prior to performing any study procedures.

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* Evidence of growth of pituitary adenoma or other intracranial tumor within the last 12 months (confirmed by computer tomography (CT) or magnetic resonance imaging (MRI) scan (with contrast) within 3 months prior to study entry or at screening).
* History of malignancy other than i) cranial irradiation (for cranial tumor or leukemia) causing GHD or ii) fully treated basal cell carcinoma
* Signs of intracranial hypertension at screening
* Heart insufficiency, NYHA class greater than 2
* History of impaired glucose tolerance, insulin resistance or overt diabetes mellitus defined according to the American Diabetes Association (ADA) Criteria
* Impaired liver function defined as elevation of liver enzymes >2 x upper limit of normal
* Impaired kidney function defined as increased serum creatinine levels >1.5 x upper limit of normal
* Active acromegaly in the last 18 months and less than 6 months of active r- hGH replacement therapy
* Active Carpal tunnel syndrome
* Prader-Willi syndrome
* Active Cushing's syndrome within the last 12 months
* Systemic corticosteroids other than in replacement doses within the 3 months before study entry (temporary adjustment of glucocorticoids, as appropriate, is acceptable)
* Anabolic steroids other than gonadal steroid replacement therapy within 2 months before study entry
* History of non-compliance with medications, un-cooperativeness or drug abuse
* Blood donation or any major blood loss >500 mL within the past 90 days prior to study entry
* Patients who, based on the investigator's judgment, have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Conditions may include cardiovascular, peripheral vascular, pulmonary, hepatic, renal, or neurological disease, as determined by medical history, physical examination, laboratory tests or ECG
* Patients who participated in any investigational medicinal product (IMP) study within the last 2 months
* History of positive serology to HBC, HBV and HIV

Ages: 23 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
1. Safety and Tolerability | Following 4 weeks of MOD-4023 treatment
  Adverse events (AE's), vital signs, electrocardiogram (ECG), laboratory tests, local reaction
Maintenance of normal Insulin-like-Growth-Factor-1 (IGF-1)levels in GHDA | Following 4 weeks MOD-4023 treatment
  The primary efficacy endpoint will be the mean time interval of IGF-I levels that lay within ±1.5 SDS after the last dose administration during stage I (4w treatment) expressed in hours.

SECONDARY OUTCOMES:
Change of IGF-I levels over time expressed in absolute and SDS values | Following 4 and 16 weeks of MOD-4023 treatment
Change of IGFBP-3 over time expressed in absolute values | Following 4 and 16 weeks of MOD-4023 treatment
Number of IGF-1 normalized patients in stage II | Following 16 weeks of MOD-4023 treatment
  Number of patients achieving normalization of IGF-1 levels during dose titration 16-week treatment extension

CONTACTS AND LOCATIONS:
Locations (15):
- Czechia (2):
  - Internal Clinic in University Hospital St. Anna, Brno
  - University Hospital, 2nd Department of Internal Medicine, Hradec Králové
- Hungary (6):
  - State Health Center, 2nd department of internal medicine, Budapest
  - Semmelweis University, 2nd Clinic of Internal Medicine, Budapest
  - Petz Aladár County Teaching Hospital, Department of Endocrinology, Metabolism and Diabetology, Győr
  - University of Pécs, Medical School, 1st Department of Internal Medicine, Pécs
  - Szeged University, 1st Internal Medicine Clinic, Endocrinology, Szeged
  - Hetényi Géza Hospital and Out-Patient Clinic, 1st Department of Internal Medicine, Szolnok
- Israel (2):
  - Endocrinology and Metabolism Service, Hadassah-Hebrew University Medical Center, Jerusalem
  - Institute of Endocrinology, Tel Aviv-Sourasky Medical Center, Tel Aviv
- Clinical Center of Serbia, Institute for endocrinology, diabetes and metabolism disease, Belgrade, Serbia
- Slovakia (3):
  - . Department of Internal Medicine V, University Hospital Ruzinov, Bratislava
  - Slovak Health University, Division of Endocrinology, Bratislava
  - National Institute of Endocrinology and Diabetology, Ľubochňa
- University Medical Centre Ljubljana, Department of Endocrinology, Diabetes and Metabolic Diseases, Ljubljana, Slovenia